CLINICAL TRIAL: NCT05124496
Title: Validation of the HyperDetector Digital Solution Screening Assay for Rapid Screening for Potential SARS-CoV-2 (COVID-19) Infection
Brief Title: Validation of HyperDetector for SARS-CoV-2
Status: Suspended | Type: Observational
Why Stopped: Collected sufficient samples for analysis
Sponsor: HyperSpectral APD (Industry)
Responsible Party: Sponsor
Other Study IDs: 20204146
Record Dates: First submitted 2021-11-15; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: SARS-COV2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Comparison to Rt-PCR
  Interventions: Device: Screening Device

INTERVENTIONS:
Device: Screening Device — Screening device comparing Rt-PCR positive and negative results to HyperDetector results

SUMMARY:
To evaluate the HyperDetector as a method to rapidly screen SARS-CoV-2

To determine the sensitivity and specificity of the screening assay performed on oral swab and saliva specimens, compared to a validated RT-PCR COVID-19 method using nasal or nasopharyngeal swabs and to separately collected nasal swabs, oral swabs, oral rinse and saliva samples.

To determine the best workflow for using such an assay to reflex suspicious/positive samples to a validated RT-PCR COVID-19 assay.

ELIGIBILITY:
Inclusion Criteria:

* Subjects at COVID-19 testing site for Rt-PCR test.

Exclusion Criteria:

* Minors under the age of 5

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals obtaining Rt-PCR test
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-12-11 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | By 12/30/2022
  To determine the sensitivity of the screening assay
Specificity | By 12/30/2022
  To determine the specificity of the screening assay

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Stack, Study Director — HyperSpectral APD, LLC
Locations (1):
- HyperSpectral APD, LLC, Alexandria, Virginia, United States

IPD SHARING:
Plan to Share IPD: No